CLINICAL TRIAL: NCT03776630
Title: Exploring the Potential of Novel Biomarkers Based on Plasma microRNAs for a Better Management of Pelvic Gynecologic Tumors
Acronym: GYNO-MIR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: K160922J; 2018-A00018-47 (Other: ANSM)
Record Dates: First submitted 2018-09-24; First posted 2018-12-17 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Endometrial Cancer
Keywords: Ovarian cancer; endometrial cancer; miR; diagnostic
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Patients undergoing surgery for benign pelvic lesions
  Interventions: Other: Blood sample
- Ovarian Cancer (Other)
  Interventions: Other: Blood sample
- Endometrial Cancer (Other)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Two blood samples (2 tubes of 4 ml for each blood sample) will be collected per patient during the study period for EC and OC. One blood sample will be collected for control population. The first sample will be collected prior to any treatment for EC, OC, and control population.
  For EC, the second collection will be done one month post-surgery. For OC, the second collection will be done 6 to 9 months after the initial diagnosis, in most cases at the completion of adjuvant chemotherapy. For control population, there will be no second sample.

SUMMARY:
This trial is a non-randomized, open label and multicenter study.

It aims to :

for endometrial cancer.:validate the 5-miR index assessed in plasma samples as a diagnostic marker to assess the risk of lymph node metastases for ovarian cancer : to validate the previous finding on the prognostic value of the pre-/post-treatment variation of miR200b plasma concentrations with regards to PFS (the investigators mean the primary treatment including up-front or post-chemotherapy debulking and adjuvant chemotherapy).

DETAILED DESCRIPTION:
MicroRNAs (miRs) have been linked to carcinogenesis and can act as metastatic activators or suppressors. There is now ample evidence that circulating miRs can be used as biomarkers. This project is focused on ovarian (OC) and endometrial cancers (EC), respectively the deadliest and most frequent gynecologic malignancies.

The main challenge for physicians managing women with early-stage EC is when to opt for lymphadenectomy. Tools that are currently used are not accurate enough to identify women with increased risk of nodal metastases. Ballester's team recently found a relationship between the high expression of a set of 5 miRs in the primary tumor and nodal status.

OC is the leading cause of death from gynecological cancer. The prognosis depends on the response of the residual tumor mass to adjuvant chemotherapy. Currently, this response remains largely unpredictable and even difficult to monitor with CA125 measurements and current imaging techniques. Busson's team recently showed that the variation of plasma miR200b during primary treatment is predictive of progression-free survival (PFS).

The study involves 3 populations of participants :

* Patients with EC
* Patients with OC
* Patients undergoing surgery for benign pelvic lesions (control population)

ELIGIBILITY:
Inclusion Criteria:

For all patients (EC, OC, Control)

* Written informed consent;
* Age ≥ 18 years old;
* Patient affiliated to social security.

EC patients

* Histologically proven EC ;
* Type 1 and 2 EC;
* FIGO stage I or II or III EC requiring first intention surgical staging.

OC patients

* Histologically proven OC or strong suspicion of OC on clinical arguments (abdomino-pelvian mass detected by palpation or echography and/or ascitis and/or elevated CA125);
* Epithelial OC: any histological subtype;
* FIGO stage I to IV OC.

Control patients - Any lesion which is supposed to be benign and requires surgery. -

Exclusion Criteria:

For all patients (OC, EC, Control)

* Unable or unwilling to comply with the protocol requirements and/or unwilling to sign an informed consent form.
* Deprived of liberty or under legal protection measure;
* Ongoing pregnancy;

Control patients:

- Previous history of cancer.

EC patients

* FIGO stage IV at preoperative imaging techniques.
* Previous history of cancer. OC patients
* Non epithelial cancer.
* Previous history of cancer - except for patients who developed breast cancer at least 5 years or more before ovarian cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
For EC: presence or absence of lymph-node metastases according to pathological analysis (reference technique). | 2 months
  To validate the 5-miR index assessed in plasma samples as a diagnostic marker to assess the risk of lymph node metastases.
For OC: PFS or death for any cause at 24 months. | 24 months
  To validate the previous finding on the prognostic value of the pre-/post-treatment variation of miR200b plasma concentrations with regards to PFS (by OC treatment, we mean the primary treatment including up-front or post-chemotherapy debulking and adjuvant chemotherapy).

SECONDARY OUTCOMES:
It aims to investigate the links of the 5-miR index with classical predictors of lymph node involvement in the context of EC. | 2 months
  Histopathological characteristics of the tumor in the context of EC: grade
It aims to investigate the links of the 5-miR index with classical predictors of lymph node involvement in the context of EC (1) | 2 months
  Histopathological characteristics of the tumor in the context of EC: type endometrioid vs. non endometrioid
It aims to assess the prognostic value of pre/post-operative plasma miR variations in terms of PFS in EC and OC | 60 months
  PFS for both EC and OC
It aims to assess the prognostic value of pre/post-operative plasma miR variations in terms of OS in EC and OC | 60 months
  OS (defined as the time from the start of the treatment to death) for both EC and OC
Sensitivity and specificity of plasma miR detection by RCA-FRET applied directly on plasma samples or following RNA extraction. | 60 months
  it aims to validate multiplexed homogenous miR detection based on RCA-FRET compared to conventional qRT-PCR in plasma samples. It also aims to search for novel plasma miRs potentially informative on lymph node involvement (EC) or PFS (OC) by high throughput sequencing (RNA seq).

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy CANLORBE, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de chirurgie et oncologie gynécologique et mammaire, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided